CLINICAL TRIAL: NCT01901315
Title: New Information and Communication Technologies in the Delivery of Mental Health Treatment: Psychiatric Care Via Videoconferencing
Brief Title: Psychiatric Care Via Videoconferencing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IPQ-0782/11
Record Dates: First submitted 2013-07-10; First posted 2013-07-17 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2013-07

CONDITIONS: Depression
Keywords: telepsychiatry; telemental health; teleassistance; health care delivery; depression; Telemedicine; Remote Consultation; Videoconferencing; Community Mental Health Services
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Online consultation (Experimental): Monthly video consultations with psychiatrist
  Interventions: Procedure: Online consultation
- Face-to-face consultation (Experimental): Monthly face-to-face consultations with psychiatrist
  Interventions: Procedure: Face-to-face consultation

INTERVENTIONS:
Procedure: Online consultation — Patients in the online consultation (intervention) group have monthly consultation with their attending psychiatrist through videoconferencing during one year. After each consultation, the medication is sent to the patient through a home delivery program. For reasons of patient safety, consultations at baseline, and after 6 and 12 months will be realized in a face-to-face form at the Institute of Psychiatry (IPq).
  Arms: Online consultation
Procedure: Face-to-face consultation — Patients in the face-to-face consultation (control) group have monthly face-to-face consultation with their attending psychiatrist during one year at the Institute of Psychiatry (IPq).
  Arms: Face-to-face consultation

SUMMARY:
The purpose of this project is to compare the effectiveness between face-to-face consultations and consultations via videoconferencing among patients treated in the Institute of Psychiatry (IPq).

DETAILED DESCRIPTION:
Introduction: Within the emergence of the Internet and for the purposes of providing psychiatric services across distances, the provision of mental health service via video counseling has become a possible way of mental health service delivery. An appropriate systematization of the propaedeutic methods in psychiatry, according to the interactive resources of telemedicine, and a standardized assessment based on clinical records turn this method to a viable alternative for service delivery all over the world. The main benefit of video counseling is an increased access to care services. But, so far, there is still limited research regarding to the effectiveness of telepsychiatry in the management of mental illnesses.

Objective: To verify the applicability of psychiatric attendance via Interned-based videoconferencing, comparing various quality characteristics between this method and face-to-face attendance, on the basis of a one-year follow-up study with a randomized clinical trial (RCT) design.

Material and methods: 100 patients of the Institute of Psychiatry (IPq) between 18 to 55 years old with depressive disorders are randomly allocated to a control (monthly face-to-face consultation with the attending psychiatrist) or intervention group. The intervention group will have consultations with the attending psychiatrist through internet-based videoconference. For reasons of patient safety, consultations at baseline, and after 6 and 12 months will be realized in a face-to-face form for all patients. At baseline, and after 6 and 12 months mental health, satisfaction with treatment, therapeutic relationship, and medical compliance will be assessed. Depression will be assessed at baseline, and after 3, 6, 9 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* depressive disorder
* between 18 to 55 years
* broadband Internet access

Exclusion Criteria:

* Hamilton Depression Rating Scale total score > 15
* severe cognitive limitations

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2012-03; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Baseline Depression Severity | 0 months (baseline)
  Instrument: Hamilton Depression Rating Scale
Change from Baseline in Depression Severity at 6 months | 6 months
  Instrument: Hamilton Depression Rating Scale
Change from Baseline and 6-months Follow-up in Depression Severity at 12 months | 12 months
  Instrument: Hamilton Depression Rating Scale
Baseline Satisfaction with Treatment | 0 months (baseline)
  Instrument: Client Satisfaction Questionnaire (CSQ-8)
Change from Baseline in Satisfaction with Treatment at 6 months | 6 months
  Instrument: Client Satisfaction Questionnaire (CSQ-8)
Change from Baseline and 6-months Follow-up in Satisfaction with Treatment at 12 months | 12 months
  Instrument: Client Satisfaction Questionnaire (CSQ-8)
Baseline Mental Health | 0 months (baseline)
  Instrument: Mental Health Inventory (MHI)
Change from Baseline in Mental Health at 6 months | 6 months
  Instrument: Mental Health Inventory (MHI)
Change from Baseline and 6-months Follow-up in Mental Health at 12 months | 12 months
  Instrument: Mental Health Inventory (MHI)
Baseline Quality of Therapeutic Relationship | 0 months (baseline)
  Instrument: Working Alliance Inventory (WAI)
Change from Baseline in Quality of Therapeutic Relationship at 6 months | 6 months
  Instrument: Working Alliance Inventory (WAI)
Change from Baseline and 6-months Follow-up in Quality of Therapeutic Relationship at 12 months | 12 months
  Instrument: Working Alliance Inventory (WAI)
Baseline Medical Adherence | 0 months (baseline)
  Instrument: self-reported measure of medication adherence with four items:
  * Do you forget to take your medication?
  * Are you careless at times about taking your medicine?
  * When you feel better, do you sometimes stop taking your medicine?
  * Sometimes when you feel worse, do you stop taking your medicine?
  Response categories are yes/no for each item with a dichotomous response and a 5-point Likert response for the last item.
Change from Baseline in Medical Adherence at 6 months | 6 months
  Instrument: self-reported measure of medication adherence with four items:
  * Do you forget to take your medication?
  * Are you careless at times about taking your medicine?
  * When you feel better, do you sometimes stop taking your medicine?
  * Sometimes when you feel worse, do you stop taking your medicine?
  Response categories are yes/no for each item with a dichotomous response and a 5-point Likert response for the last item.
Change from Baseline and 6-months Follow-up in Medical Adherence at 12 months | 12 months
  Instrument: self-reported measure of medication adherence with four items:
  * Do you forget to take your medication?
  * Are you careless at times about taking your medicine?
  * When you feel better, do you sometimes stop taking your medicine?
  * Sometimes when you feel worse, do you stop taking your medicine?
  Response categories are yes/no for each item with a dichotomous response and a 5-point Likert response for the last item.

OTHER OUTCOMES:
Demographics | 0 months (baseline)
  Age, Gender, Nationality, Marital Satus, Education, and Employment
Technical Control of Online Consultations at 6 an 12 months | 6 and 12 months
  Assessment of technical aspects regarding to online consultations: sound quality, video quality, speed, technical support

CONTACTS AND LOCATIONS:
Overall Officials: Wagner F Gattaz, Prof. Dr., Study Director — Institute of Psychiatry (IPq)
Locations (1):
- Institute of Psychiatry, School of Medicine, University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Hungerbuehler I, Valiengo L, Loch AA, Rossler W, Gattaz WF. Home-Based Psychiatric Outpatient Care Through Videoconferencing for Depression: A Randomized Controlled Follow-Up Trial. JMIR Ment Health. 2016 Aug 3;3(3):e36. doi: 10.2196/mental.5675. PMID 27489204